CLINICAL TRIAL: NCT04128995
Title: Surgical or Medical Treatment for Pediatric Type 2 Diabetes
Brief Title: Surgical or Medical Treatment
Acronym: ST2OMP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Amy Shah, Professor, Department of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK119450 (NIH)
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 2; Pediatric Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Open label prospective clinical trial. Primary comparison is medical (n=45) vs surgical (n=45) groups. Patients with obesity and no diabetes (n=10) are a comparator group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Medical Therapy and Bariatric Surgery in Youth with Type 2 Diabetes (Active Comparator): Youth with type 2 diabetes undergoing bariatric surgery, n=45
  Interventions: Procedure: Advanced Medical Therapy and Bariatric Surgery
- Medical Therapy in Youth with Type 2 Diabetesin Youth with Type 2 Diabetes (Active Comparator): Youth with type 2 diabetes receiving medical management, n=45
  Interventions: Drug: Advanced Medical Therapy
- Bariatric Surgery in Youth with Obesity (Active Comparator): Youth with no obesity undergoing bariatric surgery, n=10
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Advanced Medical Therapy and Bariatric Surgery — Vertical Sleeve Gastrectomy and Advanced Medical Therapy that could include metformin, GLP-1 agonist, SGLT-2 inhibitor, or basal insulin for youth with type 2 diabetes
  Arms: Medical Therapy and Bariatric Surgery in Youth with Type 2 Diabetes
Drug: Advanced Medical Therapy — Advanced Medical Therapy that could include metformin, GLP-1 agonist, SGLT-2 inhibitor, or basal insulin for youth with type 2 diabetes
  Arms: Medical Therapy in Youth with Type 2 Diabetesin Youth with Type 2 Diabetes
Procedure: Bariatric Surgery — Vertical Sleeve Gastrectomy for youth without type 2 diabetes
  Other Names: Vertical Sleeve Gastrectomy
  Arms: Bariatric Surgery in Youth with Obesity

SUMMARY:
This study will test the hypothesis that metabolic bariatric surgery will be more effective at providing durable glycemic control and reduce co-morbidities than intensive medical therapy in youth with type 2 diabetes.

DETAILED DESCRIPTION:
Youth-onset type 2 diabetes (T2D) leads to early dependence on exogenous insulin and progression of T2D co-morbidities, including dyslipidemia, hypertension, non-alcoholic fatty liver disease and diabetic kidney disease. The pathophysiology of T2D in youth differs considerably from adults and current treatment approaches are in-adequate for youth. Thus, exploration of innovative approaches to reduce co-morbidities is critical. Metabolic bariatric surgery (MBS) significantly improves multiple outcomes in adults with T2D. Initial small, uncontrolled studies of Roux-en-Y gastric bypass also suggest beneficial effects in youth with T2D, but definitive studies and understanding of mechanisms in youth-onset T2D are lacking, especially with the now more common form of MBS, vertical sleeve gastrectomy (VSG).

We will test the hypothesis that VSG will be more effective in reducing glycemia and comorbidities than the best currently available medical treatment: advanced medical therapy (AMT), via pancreatic, enterohepatic and/or metabolic changes. To test this hypothesis, 90 adolescents with T2D will be studied to compare the effects of VSG vs. AMT on glycemic control and T2D-associated comorbidities, as well as underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria for the medical or surgical type 2 diabetes groups

* Age 13-19.9 years of age at time of signing the consent
* Type 2 diabetes by the American Diabetes Association criteria
* Negative diabetes-associated antibodies

Exclusion Criteria for the medical or surgical type 2 diabetes groups Known type 1 diabetes, maturity onset diabetes of the young (MODY), or secondary diabetes

* Any chronic oral steroids use within 60 days of enrollment
* Current pancreatotoxic drugs
* Chronic kidney or liver disease (except NAFLD or DKD)
* Pregnancy, breast-feeding or intension of becoming pregnant
* Prior bariatric surgery
* History of malignancy
* Current participation in another clinical trial that may affect study outcomes
* Other conditions, that in the determination of the study investigator, may interfere with study participation
* Inclusion Criteria for the Obese control group
* Age 13-19.9 years of age at time of signing the consent
* Clinical indication to receive bariatric surgery

Exclusion Criteria for the obese control group

* Known diabetes
* Any chronic oral steroids use within 60 days of enrollment
* Current pancreatotoxic drugs
* Chronic kidney or liver disease (except NAFLD or DKD)
* Pregnancy, breast-feeding or intension of becoming pregnant
* Prior bariatric surgery
* History of malignancy
* Current participation in another clinical trial that may affect study outcomes
* Other conditions, that in the determination of the study investigator, may interfere with study participation

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | At one year
  Hemoglobin A1c of <6.5%

SECONDARY OUTCOMES:
Glycemic Control | At two years
  Hemoglobin A1c <6.5% at 2 years
Glycemic Variability | At one year
  Time In Range by Continuous Glucose Monitoring
Beta Cell Function | at 1 and 2 years
  Oral disposition index= Insulin secretion [insulinogenic index] * insulin sensitivity [1/fasting insulin]
Alpha cell function | at 1 and 2 years
  Glucagon area under the curve from mixed meal tolerance testing
Incretin Response | at 1 and 2 years
  GLP-1 area under the curve from mixed meal tolerance testing
Fatty Liver Disease | at 1 and 2 years
  Hepatic Fat (<5% )by Magnetic Resonance imaging
Dyslipidemia | at 1 and 2 years
  LDL <130mg/dL
Hypertension | at 1 and 2 years
  Blood pressure <130/80 mmHg
Diabetic Kidney Disease | At 1 and 2 years
  Urinary albumin excretion <30μg/mg

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Shah, MD MS, Principal Investigator — Cincinnati Childrens Hospital Medical Center; Kristen J Nadeau, MD MS, Principal Investigator — Children's Hospital Colorado; Michael A Helmrath, MD MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Thomas H Inge, MD PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Lurie Children's Hospital, Chicago, Illinois
  - Cincinnati Childrens, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
The PI's will also report a of summary results information (including adverse events) after completion of the study. All data from the study including any negative findings will be published in peer reviewed manuscripts.

REFERENCES:
- [Derived] Shah AS, Helmrath MA, Inge TH, Xanthakos SA, Kelsey MM, Jenkins T, Trout AT, Browne L, Nadeau KJ. Study protocol: a prospective controlled clinical trial to assess surgical or medical treatment for paediatric type 2 diabetes (ST2OMP). BMJ Open. 2021 Aug 13;11(8):e047766. doi: 10.1136/bmjopen-2020-047766. PMID 34389568